CLINICAL TRIAL: NCT05921188
Title: Identification of Treatment Parameters That Maximize Language Treatment Efficacy for Children
Brief Title: The Effect of Prior Learning on Word Learning
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Late Talker Phase 4; 2R01DC015642-06 (NIH)
Record Dates: First submitted 2023-06-14; First posted 2023-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Language Development Disorders
Keywords: Late Talkers
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Intervention Model Description: The investigators will use treatment effect sizes to compare children to themselves (treatment v. control) and across groups (More Familiar Sounds v. Less Familiar Sounds).
Who Masked: Participant, Care Provider
Masking Description: The children in the study and their caregivers will not be told which treatment group their child is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- More Familiar Sounds (Experimental): Children in this condition will learn new words whose sounds are more like the sounds in the words the child already understands.
  Interventions: Behavioral: VAULT Phase 4
- Less Familiar Sounds (Active Comparator): Children in this condition will learn new words whose sounds are less like the sounds in the words the child already understands.
  Interventions: Behavioral: VAULT Phase 4

INTERVENTIONS:
Behavioral: VAULT Phase 4 — Children will receive an input-based word learning treatment that is designed based on principles of statistical learning.

SUMMARY:
The goal of this clinical trial is to compare two treatment conditions for late talking toddlers. In 8 weeks of word learning treatment, toddlers will be taught words that sound more like the words they already know or sound less like the words they already know. The investigators see which group learns more, to understand if choosing words that let children use the knowledge they already have helps with learning.

DETAILED DESCRIPTION:
Late talking toddlers will be assigned to be in the More Familiar Sounds condition or the Less Familiar Sounds condition. Both groups will receive 8 weeks of Vocabulary Acquisition and Usage for Late Talkers (VAULT) word learning treatment (2x/week for 30 minutes per session) using their words. The investigators will compare learning within children (taught words v. control words that are not explicitly taught) to make sure the learning that is happening is due to the treatment and not just maturation. The investigators will compare across groups to see if the group treated with More Familiar Sounding words learns more than the group treated with Less Familiar Sounding words.

ELIGIBILITY:
Inclusion Criteria:

* Native English Speaking
* Pass pure tone hearing screening or medical report of normal hearing
* 2-3 Years of age at start of study
* MCDI expressive scales <10th percentile

Exclusion Criteria:

* Parental reports of other diagnoses
* Enrolled in concurrent treatment elsewhere
* Nonverbal IQ <75 as measured by the Bayley scales
* Parents unable to consistently bring child to treatment sessions

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Treatment Effect Size | Change from baseline through treatment, which will average an 8-week time frame.
  The investigators will count the number of spontaneous and probed productions of target and control words and calculate a treatment effect size (d).
Number/Rate of Words Learned | Change from Initial Evaluation through Follow-up, which will average a 6-month time frame.
  The investigators will measure the number of words learned and the rate of words learned as reported by the parent on the MCDI starting prior to treatment and measured during, immediately following, and 4-6 weeks after the treatment.

SECONDARY OUTCOMES:
Post Treatment Retention | Change from end of treatment to follow up, which will average 4-6 weeks.
  The investigators will use probe data and parental report to determine how many of the words the child retained from treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Alt, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No